CLINICAL TRIAL: NCT01899703
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Repeat Doses of GSK2330672 Administration in Patients With Primary Biliary Cirrhosis (PBC) and Symptoms of Pruritus
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Repeat Doses of GSK2330672 Administration in Subjects With Primary Biliary Cirrhosis (PBC) and Symptoms of Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 117213
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cholestasis, Intrahepatic
Keywords: Intestinal bile acid transport inhibitor; Pruritus; Primary biliary cirrhosis; Ursodeoxycholic acid; GSK2330672; Pharmacokinetics
MeSH Terms: conditions — Cholestasis, Intrahepatic; Pruritus; Liver Cirrhosis, Biliary | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2330672 (Experimental): Subject will receive GSK2330672 45 mg BID from Day 1 to 3 and 90 mg BID from Day 4 to 14 of one of the two treatment periods. Patients were randomized to one of two sequences receiving either (i) GSK2330672 followed by placebo; OR (ii) placebo followed by GSK2330672.
  Interventions: Drug: GSK2330672; Drug: Placebo; Drug: Ursodeoxycholic acid
- Placebo (Experimental): Subject will receive placebo BID from Day 1 to 14 of one of the two treatment periods. Patients were randomized to one of two sequences receiving either GSK2330672 followed by placebo; OR placebo followed by GSK2330672.
  Interventions: Drug: GSK2330672; Drug: Placebo; Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: GSK2330672 — GSK2330672 oral preserved solution 1.5mg/g will be supplied in amber glass bottles and as per randomization schedule subject will receive 45 mg BID from Day 1 to 3 and 90 mg BID from Day 4 to 14 of one of the two treatment periods.
Drug: Placebo — Placebo oral preserved solution will be supplied in amber glass bottles and as per randomization schedule subject will receive placebo BID from Day 1 to 14 of one of the two treatment periods. .
Drug: Ursodeoxycholic acid — UDCA 250 mg will be supplied in capsule form. The subjects, who are taking UDCA at the time of Run-in-period, will be continued on the same total daily dose of drug but converted to a standardized formulation and a standardized dosing regimen administering the entire daily dose once daily in the evening before bedtime. Once daily dosing of UDCA will continue for the duration of the study.

SUMMARY:
This will be a randomized, double-blind, placebo-controlled study to assess safety and tolerability of GSK2330672 administration in subjects with primary biliary cirrhosis (PBC) and symptoms of pruritus. It is a double-blind, crossover study with subjects receiving placebo or GSK23306772 in random order during two 14-day treatment periods. Additionally, the study will determine GSK2330672 exposure and interactions with ursodeoxycholic acid (UDCA). The total duration of subject participation will be 14 weeks for screening (45 days) and the treatment period. Subjects who are eligible for enrolment will participate in a 2-week placebo run-in period. Subjects will be randomized in a crossover fashion (Sequence 1 / Sequence 2) to receive placebo or GSK2330672 treatment during two consecutive 2-week study periods. Subjects will then participate in a 2-week placebo dosing follow-up period ending in final follow-up assessments. Study results will be utilized to form a benefit: risk profile for GSK2330672 in PBC that will determine plans for progression to exploratory efficacy trials

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Proven or likely PBC, as demonstrated by the subject presenting with at least 2 of the following: history of sustained increased alkaline phosphatise (AP) levels first recognized at least 6 months prior to Day 1; positive antimitochondrial antibodies (AMA) titer (>1:40 titer on immunofluorescence or M2 positive by enzyme-linked immunosorbent assay [ELISA]) or PBC-specific antinuclear antibodies (antinuclear dot and nuclear rim positive); liver biopsy consistent with PBC.
* Screening AP value between <=<10 × upper limit of normal (ULN).
* Subjects should be on stable doses of UDCA for >8 weeks at time of screening. Subjects not taking UDCA due to intolerance may be enrolled into this study following agreement by the GSK medical monitor.
* Symptoms of pruritus as follows (one of the following): PBC subjects with severe symptoms of pruritus that significantly impact daily life and have proven refractory after at least one previous therapy has been discontinued due to inadequate clinical response, poor tolerability or adverse events. Temporary response to cooling, 1% menthol in aqueous cream, nasobiliary drainage or molecular adsorbent recirculating system (MARS) therapy is still compatible with refractory itch; PBC subjects with unresolved symptoms with use of a single antipruritic agent who can tolerate washout of current therapy for the duration of the trial; PBC subjects seeking treatment for pruritus that is newly diagnosed or previously untreated.
* A female subject is eligible to participate if she is not pregnant, as confirmed by a negative serum human chorionic gonadotrophin (hCG) test or at least one of the following conditions applies: Non-reproductive potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli-international units per milliliter and estradiol <40 picograms per milliliter (<147 picomole per liter) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods along with either a second form of highly effective contraception or barrier protection (condoms with spermicide) if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment; Reproductive potential and agrees to follow one of the contraception options methods for the specified duration of time.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Screening total bilirubin >1.5x ULN. Isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%.
* Screening alanine aminotransferase or aspartate aminotransferase >4x ULN.
* Screening serum creatinine >2.5 milligrams per decilitre (221 micromole/liter).
* History or presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy, or poorly controlled ascites).
* History or presence of other concomitant liver diseases including hepatitis due to hepatitis B or C virus (HCV, HBV) infection, primary sclerosing cholangitis (PSC), alcoholic liver disease, definite autoimmune hepatitis or biopsy proven nonalcoholic steatohepatitis (NASH).
* Administration of the following drugs at any time during the 3 months prior to screening for the study: colchicine, methotrexate, azathioprine, or systemic corticosteroids.
* Current or chronic history of inflammatory bowel disease, chronic diarrhea, Crohn's disease or diarrhea related to malabsorption syndromes.
* Fecal occult blood positive test at screening.
* Based on averaged corrected QT interval (QTc) values of triplicate ECGs obtained at least 5 minutes apart: QTc >=450 milliseconds (msec); or QTc >=480 msec in subjects with Bundle Branch Block.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with any on-treatment adverse event (AE) or serious adverse event (SAE) from Baseline to Day 56 | Up to Day 56
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, important medical events which may require medical or surgical interventions.
Change from Baseline in white blood cell count (WBC), total neutrophil, lymphocyte, monocyte, eosinophil, basophil, and platelet counts at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  White blood cell, total neutrophil, lymphocyte, monocyte, eosinophil, basophil, and platelet counts were measured at Baseline, Day 28 (D28), Day 42 (D42) and Follow-up (Day 56). Change from baseline is summarized for these parameters. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the baseline visit, the last pre-dose value at the baseline visit was considered as baseline. Change from baseline was calculated as Post-Baseline Visit value minus Baseline values.
Change from Baseline in hemoglobin and mean corpuscle hemoglobin concentration (MCHC) at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  Hemoglobin and MCHC were measured at Baseline, Day 28 (D28), Day 42 (D42) and Follow-up (Day 56). Change from baseline is summarized for these parameters. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the baseline visit, the last pre-dose value at the baseline visit was considered as baseline. Change from baseline was calculated as Post-Baseline Visit value minus Baseline values.
Change from Baseline in mean corpuscle volume (MCV) at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  Hematology parameters were measured at Baseline, Day 28 (D28), Day 42 (D42) and Follow-up (Day 56). Change from baseline in MCV is summarized. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the baseline visit, the last pre-dose value at the baseline visit was considered as baseline. Change from baseline was calculated as Post-Baseline Visit value minus Baseline values.
Change from Baseline in hematocrit at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  Hematology parameters were measured at Baseline, Day 28 (D28), Day 42 (D42) and Follow-up (Day 56). Change from baseline in hematocrit is summarized. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the baseline visit, the last pre-dose value at the baseline visit was considered as baseline. Change from baseline was calculated as Post-Baseline Visit value minus Baseline values.
Change from Baseline in red blood cells (RBC) and reticulocytes at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  White and red blood cell, reticulocytes, total neutrophil, lymphocyte, monocyte, eosinophil, basophil, and platelet counts, hematocrit, hemoglobin, mean corpuscle hemoglobin concentration, mean corpuscle volume were measured at Baseline, Day 28 (D28), Day 42 (D42) and Follow-up (Day 56). Change from baseline for these parameters is summarized. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the baseline visit, the last pre-dose value at the baseline visit was considered as baseline. Change from baseline was calculated as Post-Baseline Visit value minus Baseline values.
Change from Baseline in alkaline phopshatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and gamma glutamyl transferase (GGT) at Day 28, Day 42 and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  Blood samples were collected for the measurement of ALP, ALT, AST, and GGT at Baseline, Day 28 (D28), Day 42 (D42) and Follow-up (Day 56). The Baseline value was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Change from Baseline in direct and total bilirubin, creatinine, and uric acid at Day 28, Day 42 and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  Blood samples were collected for the measurement of direct and total bilirubin, creatinine, and uric acid at Baseline, Day 28 (D28), Day 42 (D42), and Follow-up (F/U) (Day 56). The Baseline value was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Change from Baseline in calcium, chloride, carbon dioxide (CO2) content/bicarbonate, glucose, potassium, sodium, and urea/blood urea nitrogen (BUN) at Day 28, Day 42 and Follow-up (Day 56) | Baseline, Day 28, Day 42 and Follow-up (Day 56)
  Blood samples were collected for the measurement of calcium, chloride, carbon dioxide content/bicarbonate, glucose, potassium, sodium, and urea/BUN at Baseline, Day 28 (D28), Day 42 (D42), and Follow-up (D56). The Baseline value was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Change from Baseline in albumin and total protein at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42, and Follow-up (Day 56)
  Blood samples were collected for the measurement of albumin and total protein at Baseline, Day 28 (D28), Day 42 (D42), and Follow-up (Day 56). The Baseline value was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Change from Baseline in urine pH at Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 28, Day 42, and Follow-up (Day 56)
  Urine samples were collected at Baseline, Day 28 (D28), Day 42 (D42), and Follow-up (Day 56). The Baseline value was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline. Change from baseline was calculated as Post-Baseline Visit value minus Baseline values.
Change from Baseline in electrocardiogram (ECG) parameters at Day 1, Day 14, Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 1, Day 14, Day 28, Day 42, and Follow-up (Day 56)
  A 12-lead ECG measurement was obtained following 10 minutes rest in semi-supine position at Baseline, Day 1 and Day 14 (Run-in period), Day 28, Day 42, and Follow-up (Day 56). Parameters included: PR interval, QRS interval, Corrected QT (QTc) and uncorrected QT intervals were analyzed. Baseline is the average of the triplicate readings taken pre-dose for the first dose. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Change from Baseline in heart rate (HR) at Day 14, Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 14 (Run-in Period), Day 28 (Period 1), Day 42 (Period 2), and Follow-up (Day 56)
  HR was measured at the following time points: Baseline, Day 14 (D14, Run-in Period), Day 28 (D28, Period 1), Day 42 (D42, Period 2) and Follow-up (Day 56). Heart rate was obtained in a semi-supine position, after 10 minutes of rest. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Change from Baseline in diastolic blood pressure (DBP) and systolic blood pressure (SBP) at Day 14, Day 28, Day 42, and Follow-up (Day 56) | Baseline, Day 14 (Run-in Period), Day 28 (Period 1), Day 42 (Period 2), and Follow-up (Day 56)
  Diastolic blood pressure and systolic blood pressure were measured at Baseline, Day 14 (D14; Run-in Period), Day 28 (D28; Period 1), Day 42 (D42; Period 2) and Follow-up (Day 56). All measurements were made in semi-supine position, after a 10-minute rest. Baseline was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit were considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Summary of responses to gastrointestinal symptom response system (GSRS) by dimension at Day 1, Day 13, Day 27, Day 41, and Follow-up (Day 56) | Day 1 and Day 13 (Run-in Period), Day 27 (Period 1), Day 41 (Period 2), and Follow-up (Day 56)
  Gastrointestinal symptom response system is a rating scale was used to assess participant-reported symptoms over the preceding 5 to 7 days. Baseline was considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit were considered as Baseline.
Fecal Occult blood testing on Day 14, Day 28, Day 42 and Follow-up (Day 56) | Day 14, Day 28, Day 42 and Follow-up (Day 56)
  Fecal occult blood monitoring was done on Day 14, Day 28, Day 42 and Follow-up (Day 56). It was a monitoring system (in form of a card) to detect symptomatic or visible gastrotintestinal bleeding or asymptomatic occult bleeding in participants. Baseline is considered to be the participant's last non-missing assessment prior to dosing. If assessments were performed more than once at the Baseline visit, the last pre-dose value at the Baseline visit was considered as Baseline.

SECONDARY OUTCOMES:
Area under curve (AUC) of serum profiles of total bile acid concentrations (T-bile acid) at Day 14, Day 28, and Day 42 | Pre-dose, and at 2 and 5 hour (h) post-dose on Days 14, 28 and 42
  Serum samples were collected on Days 14, 28 and 42 for T bile acid. Area under the curve (AUC) over the given time interval was obtained using the repeated measures Analysis of covariance (ANCOVA) analysis.
AUC of serum profiles of 7-alpha hydroxy 4-cholesten-3-one (C4) at Day 14, Day 28, and Day 42 | Pre-dose, and at 2 and 5 hr post-dose on Days 14, 28 and 42
  Serum samples were collected on Days 14, 28 and 42 for C4. AUC over the given time interval was obtained using the repeated measures ANCOVA analysis.
Summary of derived trimmed mean participant-reported itch Scores on the Pruritus 0-10 point scale (Itch type: Worst, Intensity, Bothersome and Interference) | From Day 1 to Day 56
  A 0 to 10 point scale was implemented to measure symptoms of itching as well as other associated symptoms twice daily in the morning and evening (approximately the time of drug dosing). Participants were provided with a paper or electronic diary and were asked to score the severity of their itching symptoms from "0" for no itching to "10" for the worst possible itching. Itch type Worst, Intensity, Bothersome and Interference are reported.
Summary of Participant-reported Itch scores on the 5-D Itch scale (Domain=Degree, Direction, Disability, Distribution, Duration and Overall) on Day 1, Day 13, Day 27, Day 41 and Follow-up (Day 56) | Day 1 and Day 13 (Run-in Period), Day 27 (Period 1), Day 41 (Period 2) and Follow-up (Day 56)
  The 5-D itch scale covers five dimensions of itching experienced by participants including duration, degree, direction, disability and distribution. It was reported on Day 1 and Day 13 (Run-in Period), Day 27 (Period 1), Day 41 (Period 2) and Follow-up (Day 56). The scores of each of the five domains were achieved separately and then summed together to obtain a total 5-D score. 5-D scores potentially ranged between 5 (no pruritus) and 25 (most severe pruritus).
Participant reported outcome for primary biliary cirrhosis (PBC)-40 Quality of life (QOL) scale (Domain=Symptoms) on Day 1, Day 13, Day 27, Day 41 and Follow-up (Day 56) | Day 1 and Day 13 (Run-in period), Day 27 (Period 1), Day 41 (Period 2) and Follow-up (Day 56)
  PBC-40 scale includes 6 domains (cognitive, itch, fatigue, social, emotional, and other). Symptoms with individual questions were scored between 1 to 5, a higher score indicating greater symptom and worse quality of life. The PBC-40 scale was validated for use with a 4 week recall, however, for the purposes of this study it was administered every 2 weeks on Day 1 and Day 13 (Run-in Period), Day 27 (Period 1), Day 41 (Period 2) and Follow-up (Day 56).
Dose-normalized area under the concentration-time curve (DNAUC[0-24hr]) for UDCA and its metabolites taurodeoxycholic acid (TUDCA) and glycoursodeoxcholic acid (GUDCA) on Day 14, Day 28, and Day 42 | Pre-dose and at 6, 12, 12.5, 13, 14, 15, 17, 19, 21 and 24 h on Days 14, 28 and 42
  DNAUC(0-24hr) was estimated for assessment of UDCA and its metabolites TUDCA and GUDCA. ANCOVA was used and data presented were log transformed. Blood samples were collected at following time points: pre-dose and at 6, 12, 12.5, 13, 14, 15, 17, 19, 21 and 24 h on Days 14, 28 and 42.
Dose-normalized maximum plasma concentration (DNCmax) for UDCA and its metabolites TUDCA and GUDCA on Day 14, Day 28, and Day 42 | Pre-dose and at 6, 12, 12.5, 13, 14, 15, 17, 19, 21 and 24 hours on Days 14, 28 and 42
  DNCmax was estimated for assessment of UDCA and its metabolites TUDCA and GUDCA. An analysis of variance (ANCOVA) was used and data presented were log transformed. Blood samples were collected at following time points: pre-dose and at 6, 12, 12.5, 13, 14, 15, 17, 19, 21 and 24 hours on Days 14, 28 and 42.
Plasma pharmacokinetics for GSK2330672 on Day 14, Day 28, and Day 42 | Pre-dose and post-dose 2, 10, 12 hours on Days 14, 28 and 42
  Plasma samples were collected at following time points: pre-dose and post-dose 2, 10, 12 hr on Days 14, 28 and 42. Pharmacokinetic analysis of plasma concentration-time data for these analytes were conducted using non-compartmental Model 200.
Steady state maximum plasma concentration (Cmax) for ursodeoxycholic acid (UDCA) and its metabolites taurodeoxycholic acid (TUDCA) and glycoursodeoxcholic acid (GUDCA) | Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2).
  Approximately 2 mL of whole blood was collected for UDCA and it's metabolites PK analysis at Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2). Blood sampling for UDCA and it's metabolites PK analysis was only performed in participants who were administering UDCA.
Steady state time to Cmax (Tmax) for UDCA, TUDCA, and GUDCA | Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2).
  Approximately 2 mL of whole blood was collected for UDCA and it's metabolites PK analysis at Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2). Blood sampling for UDCA and it's metabolites PK analysis was only performed in participants who were administering UDCA.
Areas under the plasma concentration-time curve(AUC)0-24hr UDCA, TUDCA and GUDCA. | Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2)
  Approximately 2 mL of whole blood was collected for UDCA and it's metabolites PK analysis at Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2). Blood sampling for UDCA and it's metabolites PK analysis was only performed in participants who were administering UDCA.
Molar Ratio of AUC(0-24) between metabolites (TUDCA and GUDCA) and parent (UDCA) | Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2).
  Approximately 2 mL of whole blood was collected for UDCA and it's metabolites PK analysis at Pre-dose (0.0, of first dose of the day), 6.0, 12.0 (Pre-dose of second dose of the day), 12.5, 13.0, 14.0, 15.0, 17.0, 19.0, 21.0 and 24.0 hr on Day 14 (end of Run-in period), 28 (end of Period 1), and 42 (end of Period 2). Blood sampling for UDCA and it's metabolites PK analysis was only performed in participants who were administering UDCA.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Birmingham, West Midlands
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hegade VS, Kendrick SF, Dobbins RL, Miller SR, Thompson D, Richards D, Storey J, Dukes GE, Corrigan M, Oude Elferink RP, Beuers U, Hirschfield GM, Jones DE. Effect of ileal bile acid transporter inhibitor GSK2330672 on pruritus in primary biliary cholangitis: a double-blind, randomised, placebo-controlled, crossover, phase 2a study. Lancet. 2017 Mar 18;389(10074):1114-1123. doi: 10.1016/S0140-6736(17)30319-7. Epub 2017 Feb 8. PMID 28187915
- [Derived] Hegade VS, Kendrick SF, Dobbins RL, Miller SR, Richards D, Storey J, Dukes G, Gilchrist K, Vallow S, Alexander GJ, Corrigan M, Hirschfield GM, Jones DE. BAT117213: Ileal bile acid transporter (IBAT) inhibition as a treatment for pruritus in primary biliary cirrhosis: study protocol for a randomised controlled trial. BMC Gastroenterol. 2016 Jul 19;16(1):71. doi: 10.1186/s12876-016-0481-9. PMID 27431238
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register